CLINICAL TRIAL: NCT03350412
Title: Multiplex Genotyping of Metastatic Colorectal Cancer Patients for Precision Medicine Clinical Trials
Brief Title: Genotyping of Metastatic Colorectal Cancer Patients for Precision Medicine Clinical Trials
Acronym: FUNNEL
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Fondazione del Piemonte per l'Oncologia (Other)
Responsible Party: Sponsor
Other Study IDs: 007-IRCC-10IIS-14
Record Dates: First submitted 2017-07-18; First posted 2017-11-22 (Actual); Last update posted 2018-10-30 (Actual); Status verified 2018-10

CONDITIONS: Metastatic Colorectal Cancer
MeSH Terms: conditions — Colorectal Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood and tumor specimens
Oversight: Data Monitoring Committee: No

SUMMARY:
The goal of delivering the right drug to the right cancer patient (precision medicine) requires a detailed understanding of how genomic alterations are linked to drug response. The purpose of this study is to intercept at point-of-care a large cohort of newly diagnosed mCRC patients to determine if it is possible to obtain personalized genetic information from each subject's tumor (tissue and blood) to triage treatment choices. In case of target positivity, patients will be conveyed, whenever possible, to self-standing, independent, hypothesis-driven POC trials as soon as they exhibit resistance to standard of care treatment.

ELIGIBILITY:
Inclusion Criteria:

* Histological confirmed adenocarcinoma of the colon or rectum with metastatic disease not amenable to salvage surgery.
* Planned primary treatment at FUNNEL center or FUNNEL center referring Hospital.
* Availability of fresh tissue or a paraffin block for genotyping NOT older than 1 year.
* Age ≥18.
* ECOG PS 0-1.
* No major comorbidities that would preclude the potential enrolment of the patient in a clinical trial.
* Signed informed consent.

Exclusion Criteria:

* Symptomatic brain metastases.
* Gastro-intestinal abnormalities, inability to take oral medication, any condition affecting absorption.
* History of another neoplastic disease (except basal cell carcinoma of the skin or uterine cervix carcinoma in situ adequately treated), unless in remission for ≥ 5 years.
* No major comorbidities that would preclude the potential enrolment of the patient in a clinical trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: FUNNEL population consists of individual at least 18 years of age with newly diagnosed metastatic colorectal carcinoma at the first sign of metastasis (adjuvant relapse or first diagnosis)
Sampling Method: Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2015-10; Primary Completion 2018-12 (Estimated); Study Completion 2019-12 (Estimated)

PRIMARY OUTCOMES:
Thoroughness to report molecular profiling | 14 days from sample acquisition
  Percentage of patients with complete genotyping report produced in less than 14 days after sample acquisition.

SECONDARY OUTCOMES:
Frequence of genetic alteration included in the panel detected in 1000 consecutive mCRC | 24 months from first patient in.
  number of patients with detected genetic alteration included in the panel (mutations and/or copy number variations) over all recruited patients.
Percentage of complete data capture for treatment-related check-point events | through study completion, an average of five years

CONTACTS AND LOCATIONS:
Overall Officials: Massimo Aglietta, md, Principal Investigator — Fondazione del Piemonte per l'Oncologia
Locations (5):
- Italy (5):
  - AOU Policlinico S Orsola - Malpighi, Bologna
  - Policlinico S.Orsola Malpighi, Bologna
  - Fondazione del Piemonte per l'Oncologia, Candiolo
  - IOV - Istituto Oncologico Veneto, Padua
  - Policlinico Universitario Campus Biomedico, Roma